CLINICAL TRIAL: NCT04778332
Title: Risk Assessment, Consequences and Epidemiology of Electric Scooter Accidents Admitted to Emergency Departments.
Brief Title: Trottinettes Urgences 2019-2020
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: Trottinette19-20
Record Dates: First submitted 2021-02-18; First posted 2021-03-03 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Traumatic Injury; Accidental Injury; Alcohol Drinking; Traffic Accident; Emergencies
Keywords: Electronic Scooter; Helmet; Traumatic injury; Alcohol Drinking; Traffic Accident; Emergencies
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries; Alcohol Drinking; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study was to evaluate the risk, consequences and epidemiology of electric scooter accidents admitted to the emergency room at St. Pierre University Hospital.

This prospective observational study aims to include any patient admitted to the Adult Emergency Department of St.Pierre University Hospital Brussels following an accident related to the use of an electric scooter in order to describe and understand the epidemiology, complications and treatment of injuries associated with this means of transport.

It is intended to include all accidents occurring in the emergency room during the period from 01/06/2019 to 30/06/2020.

DETAILED DESCRIPTION:
All patients over the age of 16 years with traumatic injuries due to an accident related to the use of an electric scooter were included in the study.

Upon admission to the Emergency Department, patients over 16 years of age who accepted were included in the study. The objectives of the study were firstly to describe the context and incidence of scooter accidents, and secondly to understand the epidemiology, complications and treatment of injuries associated with this means of transport and finally, to estimate the economic impact assessed by the number of days of post-traumatic work disability, the need for access to more specialised and therefore more expensive care (operating theatre interventions, scanner-type radiological examinations or hospitalisation in intensive care units).

The data analyzed were based on :

1) the time and day of the accident, 2) the time of presentation at the hospital (same day or after the accident), 3) the mechanism of the accident, whether there were one or two people on the scooter, 4) the use or non-use of the protective helmet, 5) the influence of alcohol ; 6) the mode of arrival at the emergency room (type of ambulance or by one's own means); 7) the injury assessment, paraclinical examinations; 8) treatments; 9) hospitalization or not; 10) temporary work interruptions .

ELIGIBILITY:
Inclusion criteria:

* All patients with traumatic lesion following electric sccoter accident
* Be able to agree to participate in the study

Exclusion Criteria:

* < 16 years
* Unconscious
* Being unable to agree to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patient presenting at the ED for traumatic lesion following e-sccoter accident
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
description of traumatic injuries | during the first 24 hours.
  description of traumatic injuries based on the medical record. Categorised by severity and by anatomical localisation.
Arrival mode | Up to one year
  By ambulance or by own means
Timing of arrival | Baseline
  Immediately after the accident or delayed visit.
Accident mechanism | Baseline
  Other party ( Pedestrians hit by the scooter, accident with another) involved or not ( Loss of balance,2 drivers on the e-scooter,
alcohol | baseline up to 24 hours
  Did the driver report to being under the influence of alcohol or not
Hour of admission | Baseline up to 24 hours
  Admission between 7am-6pm; 6pm-11pm or 11pm-7am
Ownership | Baseline up to 24 hours
  E-scooter owned or rented by the patient

SECONDARY OUTCOMES:
Treatment | Up to 24 hours
  Emergency department or operative room
Paraclinical examination | Up to 24 hours
  radiography, scanner,
orientation | Up to 24 hours
  Intensive care unit, normal hospitalisation, discharge home
Cost of the treatment | Through study completion, an average of 1 year
  Ambulance, hospitalisation, treatment in the ED or operative room , temporary incapacity for work.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre YOUATOU TOWO, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHU saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
After publication all IPD will be made available through researchgate.com profile of backup investigator
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication
Access Criteria: Acces will be granted to any researcher requesting access through Researchgate.com

REFERENCES:
- [Derived] Gan-El E, Ngatchou Djomo W, Pascu Ciobanu AM, Kaufman L, Nde Djiele F, Ulrix M, Kreps B, Plumacker A, Malinverni S, Bartiaux M, Youatou Towo P. Risk assessment, consequences, and epidemiology of electric scooter accidents admitted to an emergency department: a prospective observational study. Eur J Trauma Emerg Surg. 2022 Dec;48(6):4847-4855. doi: 10.1007/s00068-022-02019-5. Epub 2022 Jun 21. PMID 35727343